CLINICAL TRIAL: NCT00873639
Title: A Prospective, Multicentre, Open Label, Non-controlled, Observational, 24-week Study in Patients Using NovoRapid® (Insulin Aspart) and Levemir® (Insulin Detemir) in a Basal-bolus Regimen for Treatment of Type 1 Diabetes Mellitus in Romania
Brief Title: Observational Study of Type 1 Diabetics Switching From Human Insulins to Modern Insulin Analogues
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3721
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin aspart; Drug: insulin detemir

INTERVENTIONS:
Drug: insulin aspart — Effectiveness and safety data collection in connection with the use of the drug NovoRapid® and Levemir® in routine clinical practice
  Other Names: NovoRapid®; ANA
Drug: insulin detemir — Effectiveness and safety data collection in connection with the use of the drug NovoRapid® and Levemir® in routine clinical practice

SUMMARY:
This trial is conducted in Europe. The aim of this observational study is to evaluate the blood glucose control (HbA1c) using NovoRapid® (insulin aspart) and Levemir® (insulin detemir) after switch from human insulins for treatment of type 1 diabetes under normal clinical practice conditions in Romania.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with type 1 diabetes who is treated with human rapid and intermediate (NPH) insulin in basal-bolus regimen

Exclusion Criteria:

* Subjects currently being treated with insulin aspart and insulin detemir
* Subjects who were previously enrolled in this study
* Subjects with a hypersensitivity to insulin aspart or to any of the excipients
* Subjects with a hypersensitivity to insulin detemir or to any of the excipients
* Women who are pregnant or have the intention of becoming pregnant within next 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 1 diabetes patients from diabetes centres who have been deemed appropriate to receive NovoRapid® and Levemir® as new treatment in basal-balus regimen and as part of routine care by the prescribing physician.
Sampling Method: Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | at 24 weeks from baseline

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c below 7.0% and below or equal to 6.5% | at 12 weeks and 24 weeks of treatment
Change in FPG (glucose variability) | at 12 weeks and 24 weeks of treatment
Change in PPG (postprandial control) | at 12 weeks and 24 weeks of treatment
Change in insulin dose and number of injections | at 12 weeks and 24 weeks of treatment
Change in body weight | at 12 weeks and 24 weeks of treatment
Change in number of hypoglycaemic events | at 12 weeks and 24 weeks of treatment
Number of adverse drug reactions (ADR) | at 12 weeks and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bucharest, Romania

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com